CLINICAL TRIAL: NCT00249561
Title: Women's Prison TC: Outcomes, Process & Economic Analysis
Brief Title: Colorado Women's TC Project
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Dr. JoAnn Y. Sacks/Principle Investigator, National Development and Research Institutes, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-14370-1; R01DA014370 (NIH); R01-14370-1
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recovery by Choice (Experimental): A modified Therapeutic Community program.
  Interventions: Behavioral: Recovery by Choice
- Intensive Outpatient Program (Active Comparator): Designed to address substance abuse and criminality, with a focus on prevention of relapse and recidivism.
  Interventions: Behavioral: The Intensive Outpatient Program (IOP)

INTERVENTIONS:
Behavioral: Recovery by Choice — The experimental condition, the modified TC, was a 6- to 9-month program located in a separate 72-bed housing unit within the prison. Inmates progressed through four program stages with upper level inmates functioning as peer mentors for newer members. The modified, comprehensive TC treatment program focused on increasing awareness and understanding of female roles and relationships as they relate to addiction and drugs used and abused, and emotional and behavioral coping skills. Program elements addressed issues of substance abuse, relapse prevention, mental health, criminal thinking and behavior, coping with trauma and abuse, and parenting skills. All treatment staff received special training related to working with women exposed to trauma and abuse, making the program "trauma informed" and "trauma sensitive."
  Arms: Recovery by Choice
Behavioral: The Intensive Outpatient Program (IOP) — The control condition, known at the prison as the Intensive Outpatient Program (IOP), was designed to address substance abuse and criminality, with a focus on prevention of relapse and recidivism. The IOP substance abuse treatment curriculum, designed for delivery over 15 weeks, consisted of a 90-hour manual-driven course (Strategies for Self-Improvement and Change, Wanburg & Milkman, 1998), which employed a cognitive behavioral format to address underlying issues of substance use/abuse and criminal behavior.
  Arms: Intensive Outpatient Program

SUMMARY:
The major aim of the project is to document and evaluate two treatments for female offenders with substance abuse problems (TC and cognitive behavioral), simultaneously studying the process of treatment, and relating treatment process to treatment outcome.

DETAILED DESCRIPTION:
The number and proportion of substance abusing women in prison have been increasing, creating a need for programs tailored to this population, and for evaluation of such programs. The specific aims of this project were: (1) to conduct a rigorous evaluation of the effectiveness of prison TC treatment for substance abusing women offenders; (2) to investigate the treatment process for the target population and to explore the relationship between the process and outcome of treatment; (3) to evaluate the cost and cost effectiveness of treatment; and (4) to assess issues in obtaining and making use of aftercare services and provide information regarding the additional contribution of aftercare treatment. The core investigation, over four years (n=600), randomly assigned female substance abusing offenders at the Denver Women's Correctional Facility to either a TC program, Recovery By Choice, the experimental (E) condition (n=300), or to a non-TC standard program, the comparison (C) condition (n=300). The study predicted better outcomes for the TC group in an intent-to-treat analysis of all study entrants. The Aim 4 supplementary study of aftercare, with no random assignment, followed program completers from E and C as they entered mandatory aftercare, choosing either TC aftercare or a non-TC treatment alternative. The research employed a prospective, longitudinal, repeated measures assessment with five points (baseline, 6-, 12-, and 18-months post-baseline) to assess standard outcome measures (e.g., drug use, crime, and employment), as well as specific measures of particular concern to female offenders (e.g., trauma and abuse). In addition to self-report data, urine toxicology and criminal record data were obtained. The study collected process data, guided by the Texas Christian University Treatment Process Model, The project contributes to a theoretical advance in our understanding of the process of treatment for women offenders in prison TCs. It advances research through a rigorous study of TC prison program effectiveness for women compared to another, routine treatment. It guides practice by delineating treatment elements for women and by examining the effectiveness of a TC program that organizes these elements. Finally, it integrates outcome and economic analysis to inform policy and planning about the effectiveness of the TC treatment under study. Perhaps most significantly, it tests TC principles and methods found effective for substance-abusing male offenders, which have been adapted for women, thereby increasing the potential utility of these strategies.

ELIGIBILITY:
Inclusion criteria:

* at least 6 months, and no more than 24 months, remaining until parole eligibility;
* a CDOC "Standardized Offender Assessment" (SOA; CDOC, 2004) score indicative of serious substance abuse problems mandating substance abuse treatment; and
* a security risk level classification of minimum, minimum-restricted, or medium (necessary to permit participation in treatment).

Exclusion criteria:

* less than 6 months, or more than 24 months, remaining until parole eligibility;
* a CDOC "Standardized Offender Assessment" (SOA; CDOC, 2004) score that is not indicative of serious substance abuse problems mandating substance abuse treatment; or
* a security risk level classification above medium.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2001-09; Primary Completion 2007-07 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Intake CTCR Baseline & Follow-Up Protocol (CTCR Protocol) | At entry
  The CTCR Protocol (CTCR, 1992) is a structured interview that was adapted from the ASI and DATAR for use in community treatment and the criminal justice system; additional versions, including Green's Trauma Scale (Green, 1996) to measure trauma and abuse, have been developed for baseline, during treatment and community follow-up with women. It assesses the following domains: socio-demographic background, substance use, psychosocial functioning, criminal justice involvement, education, employment, parenting, peer and family support, and health.
Beck Depression Inventory-II (BDI-II) | At entry
  The BDI-II (Beck, Steer, & Brown, 1996). The BDI measures three domains of depression: Somatic Depression, Cognitive Depression and Total Depression Scores, consistent with the DSM-IV criteria for depressive disorders.
Rosenberg Self-Esteem (SES) | At entry
  The SES (Rosenberg, 1965) is the most widely used global measure of self-esteem,
Symptom CheckList 90-R (SCL90-R) | At entry
  The SCL90-R (Derogatis, 1983) measures 9 domains including: somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism, providing a global index of distress: Global Severity Index (GSI).
Diagnostic Interview Survey (DIS-IV) | At entry
  The DIS-IV (Robins et al., 1995) is a structured clinical interview to generate DSM-IV lifetime and current psychiatric and substance use/abuse diagnoses.
Parenting Practices Scale (PPS) | At entry
  The PPS measures the parenting practices among parents of children under age 12.
Social Support Arizona Social Support Scale (ASSIS) | At entry
  The ASSIS (Barrera, 1980; Barrera, Sandier, & Ramsay, 1981; Stevens, Murphy, & McGrath, 2000) measures social support networks with a series of questions regarding the people who are important to the client and the number of ways they support the individual. Areas covered by the scale include: intimate interaction, material aid, advice, positive feedback, physical assistance, social participation, negative interactions, and personal characteristic of network members.
Texas Christian University Resident Evaluation of Self and Treatment (TCU-REST)
  The TCU-REST (Knight, Simpson & Chatham, 1997; Simpson & Knight, 1998) provides measures of client process and progress in treatment in the following domains: psychological functioning (including scales for self-esteem, depression, anxiety, self-efficacy, and decision-making confidence.
Client Assessment Inventory (CAI)
  The CAI (Kressel, 1998) measures client perceptions of progress and participation in TC treatment, in 14 domains: maturity, responsibility, values, drug/criminal life style, maintaining images, work attitude, social skills, cognitive skills, emotional skills, sense of well being, accepting program structure and philosophy, participating in group activities, attachment to, and investment in, the program. The latter two scales provide measures of participation and commitment.
Circumstances, Motivation and Readiness (CMR)
  The CMR assesses motivation and readiness for treatment (Circumstances 1 (external influences to enter or remain in treatment), Circumstances 2, (external influences to leave treatment), and Motivation (internal recognition of the need to change).
Cost: Drug Abuse Treatment Cost Analysis Program (DATCAP)
Service Utilization Form (SUF)
Partner Abuse Scales (PAS)
  The PAS (Hudson, 1990) consists of two matched pairs of scales, each consisting of 25 Likert type items. The Partner Abuse:
  Physical (RASPH) and the Partner Abuse: Non-Physical (PASNP) measure self-reports of physical and non-physical abuse between partners.

SECONDARY OUTCOMES:
Colorado Department of Corrections Record Information System (CDOC-RIS)
  The CDOC-RIS will be accessed to gather data on the following measures: current charge on which incarceration is based; other previous charges; current sentence; status of violent offenses; urine toxicological information on drug and alcohol use; medical information; dates of prior incarcerations; disciplinary reports; all services received while in prison; offenses committed post-release, reincarcerations, parole information (including entry into drug abuse treatment).
Biological Specimens
  In addition to the self-report interview, self-report standardized measures, and corroborating staff ratings discussed above, biological specimens (urine samples) will be collected on half of the subjects using a random sampling procedure. Urine samples test for a wide array of substances, but are valid for drug use only in the preceding 48-72 hours. Urine specimens will be collected at T1, T2, T3 and T4. The project will also use urine tests (administered selectively) that can be obtained from the CDOC-RIS.

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn Y Sacks, Ph.D., Principal Investigator — National Development and Research Institutes, Inc.
Locations (1):
- Denver Women's Correctional Facility, Denver, Colorado, United States

REFERENCES:
- [Result] Sacks JY, McKendrick K, Hamilton Z, Cleland CM, Pearson FS, Banks S. Treatment outcomes for female offenders: relationship to number of Axis I diagnoses. Behav Sci Law. 2008;26(4):413-34. doi: 10.1002/bsl.828. PMID 18683197